CLINICAL TRIAL: NCT05518396
Title: Prospective Validation of the CoDE-HF Algorithm for the Diagnosis of Acute Heart Failure
Acronym: ProVa CoDE-HF
Status: Active, not recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: DL-2021-003; MRC/CIC8/79 (Other Grant/Funding Number: MRC Confidence in Concept); RE/18/5/34216 (Other Grant/Funding Number: British Heart Foundation)
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Acute Heart Failure; Diagnosis
Keywords: Artificial Intelligence
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CoDE-HF decision support tool — We will assess the diagnostic performance of the CoDE-HF decision support tool

SUMMARY:
Acute heart failure is a life-threatening condition where the heart is suddenly unable to pump blood around the body. It can be challenging to diagnose because the symptoms often mimic other conditions. Previous studies have showed that delays in making the correct diagnosis result in worse outcomes. We therefore developed a decision-support tool called CoDE-HF that uses a computer algorithm to combine levels of a blood test called NT-proBNP with patient factors to calculate the probability of acute heart failure for an individual.

In this project, we wish to evaluate the performance of CoDE-HF in approximately 2,000 patients attending the Emergency Department with suspected acute heart failure. We will store surplus material from their blood tests to measure NT-proBNP and link information from their electronic health records with other routinely collected medical information in regional and national databases in order to evaluate this algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the Emergency Department with acute breathlessness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients presenting to the Emergency Department with acute breathlessness will be included in this study
Sampling Method: Non-Probability Sample
Enrollment: 3808 (Actual)
Dates: Start 2021-04-25 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Adjudicated diagnosis of acute heart failure | At index presentation

SECONDARY OUTCOMES:
Subsequent hospitalisation with heart failure | 3 months
All-cause death | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Cardiovascular Science, University of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
IPD can be made available to researchers upon request to the principal investigator.

REFERENCES:
- [Background] Lee KK, Doudesis D, Anwar M, Astengo F, Chenevier-Gobeaux C, Claessens YE, Wussler D, Kozhuharov N, Strebel I, Sabti Z, deFilippi C, Seliger S, Moe G, Fernando C, Bayes-Genis A, van Kimmenade RRJ, Pinto Y, Gaggin HK, Wiemer JC, Mockel M, Rutten JHW, van den Meiracker AH, Gargani L, Pugliese NR, Pemberton C, Ibrahim I, Gegenhuber A, Mueller T, Neumaier M, Behnes M, Akin I, Bombelli M, Grassi G, Nazerian P, Albano G, Bahrmann P, Newby DE, Japp AG, Tsanas A, Shah ASV, Richards AM, McMurray JJV, Mueller C, Januzzi JL, Mills NL; CoDE-HF investigators. Development and validation of a decision support tool for the diagnosis of acute heart failure: systematic review, meta-analysis, and modelling study. BMJ. 2022 Jun 13;377:e068424. doi: 10.1136/bmj-2021-068424. PMID 35697365